CLINICAL TRIAL: NCT00109265
Title: A Phase II, Multicenter, Open-Label Clinical Trial to Evaluate the Efficacy and Safety of OSI-774 in Patients With Advanced or Metastatic Breast Cancer and Disease Progression During or Following Chemotherapy
Brief Title: A Study to Evaluate Erlotinib in Patients With Advanced or Metastatic Breast Cancer During or Following Chemotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: OSI2288g; NCT00024219 (obsolete NCT alias)
Record Dates: First submitted 2005-04-26; First posted 2005-04-26 (Estimated); Last update posted 2015-07-02 (Estimated); Status verified 2013-06

CONDITIONS: Breast Cancer
Keywords: Advanced Breast Cancer; Metastatic Breast Cancer; Cancer
MeSH Terms: conditions — Breast Neoplasms; Neoplasms | interventions — Erlotinib Hydrochloride

INTERVENTIONS:
Drug: Erlotinib HCl (OSI-774)

SUMMARY:
This is a Phase II, multicenter trial of single-agent treatment with OSI 774 in patients with histologically confirmed, incurable, locally advanced or metastatic breast cancer. Patients must have measurable disease.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Women >=18 years of age
* Histologically documented, incurable, locally advanced or metastatic breast cancer
* Disease progression on or after therapy with an anthracycline, a taxane, and capecitabine (Cohort 1), or disease progression on or after therapy with at least one chemotherapy regimen for locally advanced or metastatic disease (Cohort 2)
* Measurable disease of >=2 cm (>=1 cm on spiral CT scan). Disease at previously irradiated sites is considered measurable if there is clear disease progression following radiation therapy.
* HER2 negative, HER2 unknown, or HER2 positive and disease progression following Herceptin(R) (trastuzumab) therapy
* ECOG performance status of 0 to 2
* Life expectancy of >=3 months
* Use of effective means of contraception in women of childbearing potential
* Ability to comply with study and follow-up procedures

Exclusion Criteria:

* Pleural effusions or blastic bone lesions as the only manifestations of the current metastatic breast cancer
* Other primary malignancies within 5 years except for adequately treated carcinoma in situ of the cervix or basal or squamous cell skin cancer
* Symptomatic or untreated brain metastases
* Radiotherapy, immunotherapy, hormonal therapy, or chemotherapy within 21 days prior to Day 0 (6 weeks for nitrosoureas or mitomycin); prior therapy with an agent designed to target either the EGFR or EGFR-specific tyrosine kinase activity
* INR >4.0 for patients receiving warfarin
* Cumulative anthracycline and anthracenedione exposure as follows: doxorubicin >450 mg/m, liposomal doxorubicin >550 mg/m, epirubicin >700 mg/m, or mitoxantrone >140 mg/m
* Cardiac ejection fraction (MUGA or echocardiogram) less than the local institution lower limit of normal
* Unstable systemic disease, including active infection, uncontrolled hypertension, unstable angina, congestive heart failure, or myocardial infarction within 6 months prior to Day 0, or serious cardiac arrhythmia requiring medication
* Major surgery, biopsy of a parenchymal organ, or significant traumatic injury occurring within 21 days prior to Day 0
* History of other diseases, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that might affect the interpretation of the results of the study or render the patient at high risk from treatment complications
* Abnormalities of the cornea based on history (e.g., dry eye syndrome, Sjogren's syndrome), congenital abnormality (e.g., Fuch's dystrophy), abnormal slit-lamp examination using a vital dye (e.g., fluorescein, Bengal-Rose), and/or an abnormal corneal sensitivity test (Schirmer test or similar tear production test)
* Gastrointestinal tract disease resulting in an inability to take oral medication or a requirement for IV alimentation, prior surgical procedures affecting absorption, or active peptic ulcer disease
* Pregnancy or lactation
* Any of the following abnormal baseline hematologic values: *Granulocyte count <=1500/uL; *Platelet count <100,000/uL; *Hemoglobin <9 gm/dL (transfusion permitted)
* Any of the following abnormal baseline liver function tests: *Serum bilirubin >=1.5x upper limit of normal (ULN); *Serum ALT and AST >=2.5x ULN (>5x ULN if due to liver metastases); *Alkaline phosphatase >=2.5x ULN (>4x ULN if due to liver or bone metastases)
* Other baseline laboratory values: *Serum creatinine >=1.5x ULN or creatinine clearance <=60 mL/min; *Uncontrolled hypercalcemia (>11.5 mg/dL); *Serum albumin <=3.0 g/dL

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-05; Study Completion 2002-10 (Actual)

REFERENCES:
- [Result] Dickler MN, Cobleigh MA, Miller KD, Klein PM, Winer EP. Efficacy and safety of erlotinib in patients with locally advanced or metastatic breast cancer. Breast Cancer Res Treat. 2009 May;115(1):115-21. doi: 10.1007/s10549-008-0055-9. Epub 2008 May 22. PMID 18496750